CLINICAL TRIAL: NCT05384561
Title: L'entraînement Olfactif Comme Traitement De La Dysfonction Olfactive Post COVID-19
Brief Title: Olfactory Training As a Treatment for Olfactory Dysfunction Post COVID-19
Acronym: OTTODC19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OTTODC192022JFUQTR
Record Dates: First submitted 2022-05-19; First posted 2022-05-20 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Hyposmia; COVID-19; Parosmia; Anosmia; SARS-CoV-2 Infection
Keywords: Olfactory training; Chemosensory impairments; Persistent smell impairment
MeSH Terms: conditions — Anosmia; COVID-19; Olfaction Disorders | interventions — Olfactory Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemosensory training group 1 (Experimental): For 12 weeks, morning and evening, smell four odors namely eucalyptol, phenyl ethanol, Orange, and eugenol, for a total of five minutes per session.
  Interventions: Other: Smell training
- Chemosensory training group 2 (Experimental): For 12 weeks, morning and evening, smell four odors namely coffee aroma, cheese aroma, strawberries, and limon, for a total of five minutes per session.
  Interventions: Other: Smell training

INTERVENTIONS:
Other: Smell training — For 12 weeks, morning and evening, smell four different odors or four odorless substances for a total of five minutes per session.
  Other Names: Chemosensory training group

SUMMARY:
Olfactory dysfunction is a defining symptom of COVID-19 infection. Studies have demonstrated improved olfaction in patients with post infectious olfactory dysfunction after an olfactory training (OT). The aim of this study is to assess the clinical outcomes of olfactory training (12 weeks) therapy in the treatment of persistent olfactory dysfunctions after COVID-19. Specially, we aim to compare the effectiveness of two different olfactory training (different odors).

A group will train themselves with 4 scents (rose, orange, clove and eucalyptus) and another group with 4 different scents (cheese, coffee, strawberries and lemon). Olfaction sensory evaluation will be performed by using different olfaction tests (Sniffin' Sticks and UPSIT) and complete questionnaires to assess olfactory perception and particularly parosmia and phantosmia.

DETAILED DESCRIPTION:
Patients who meet the criteria, who have agreed to participate in this research project and sign the consent form will be placed in one of the following two groups:

● Experimental group (olfactory training)

1. Initial meeting: Each participant will be asked for a session of approximately 1:30 h which will take place in a ventilated room in the laboratory of Dr. Johannes Frasnelli at UQTR. During the hour preceding this evaluation, subjects will be asked not to smoke, eat or drink anything other than water and not to wear perfume. A research assistant will be responsible for completing the various tests. During this meeting, the following tests will be done:

   * Data collection (case report form): medical and socio-demographic questionnaire that will be used for data analysis.
   * A nasal obstruction criterion scale - NOSE
   * A subjective questionnaire on the impact of OD on quality of life - sQOD-NS
   * Chemosensory Dysfunction Home Test - TMSC
   * The UPSIT 40 test
   * The Sniffin' Sticks test
   * Test to assess the manifestation of parosmia and phantosmia
   * Teaching on the olfactory rehabilitation kit and explanation of the training protocol.
2. Treatment (12 weeks): Following the initial meeting, patients can begin training:

   ■ Participants will bring their training kit with them following the olfactory evaluation.
3. Final meeting: After 12 weeks of treatment, an appointment will be scheduled with the participant. The olfactory evaluation will be done as described in the initial meeting. During the hour preceding this evaluation, subjects will be asked not to smoke, eat or drink anything other than water and not to wear perfume. A research assistant will be responsible for administering the various tests. During this meeting, the following tests will be done:

   * A subjective questionnaire on the impact of OD on quality of life - sQOD-NS
   * Chemosensory Dysfunction Home Test - TMSC
   * The UPSIT 40 test
   * The Sniffin' Sticks test
   * Test to assess the manifestation of parosmia and phantosmia

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed positive for COVID-19 with persistent olfactory dysfunction
* Willing and able to provide written informed consent
* Understand and read the French language
* Have an internet connection and a working email address

Exclusion Criteria:

* Anosmia and hyposmia pre-covid-19
* Be known chronic rhinosinusitis with or without nasal polyposis
* Have received radiotherapy or chemotherapy for Head and Neck Tumors
* Have a diagnosis of Alzheimer's, Parkinson's, multiple sclerosis or any other neurodegenerative disease 5. Have a brain tumor or ENT diagnosis 6. History of naso-sinus surgery; 7. History of traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in olfactory score on the University of Pennsylvania Identification Test (UPSIT) [ Time Frame: Measurement will be taken at time zero (pre-intervention) and 12 weeks (post-intervention) | Measurement will be taken at time zero (pre-intervention) and 12 weeks (post-intervention)
  The UPSIT includes 4 odor-impregnated booklets that contain 10 forced-choice multiple choice questions each for participants to scratch-and-sniff to identify various odors and is a commercially available test. Normosmia is defined as ≥34 for males and ≥35 for females, and a change of 4 points or more from baseline indicates a clinically meaningful result.
Changes from baseline in olfactory score on the Sniffin's Sticks test | Measurement will be taken at time zero (pre-intervention) and 12 weeks (post-intervention)
  Sniffin' Sticks test and Taste strips: Sniffin' Sticks test (Burghardt®, Wedel, Germany) is a psychophysical test. It allows semi-objective assessment of the patient's olfactory performance by means of 3 subtests: threshold test, identification test and discrimination test. The Sniffin' Sticks Olfactory Test Kits contain pen like bodies as, for example, in pens used to write on flipcharts or whiteboards.These pen-like bodies, however, contain a fibre stick which is filled with scents. For testing, the cap should be removed so the patient can smell on the tip of the pen.
n-house test for chemosensory dysfunction (TMSC) | Measurement will be taken at time zero (pre-intervention) and 12 weeks (post-intervention)
  The TMSC is a 55-item questionnaire evaluating the three chemical senses: olfaction, taste and the trigeminal sense. First, questions with a 10-point visual analog scale make a subjective self-assessment of each of the three senses. Multiple-choice questions establish the precise characteristics of the dysfunctions of each of the senses if they are present. Secondly, a psychophysical test is administered remotely using substances typical of North American cuisines. Substances are first sniffed (peanut butter, jam, vinegar, coffee) then tasted (peanut butter, jam, salt water (1 tsp/250mL), sugar water (3 tsp/250mL)). The perceived intensity of each of the substances is reported each time on a visual analogue scale of 10 points.
Parosmia and phantosmia assessment test | Measurement will be taken at time zero (pre-intervention) and 12 weeks (post-intervention)
  This test has a first part with four questions that aim to assess the presence of parosmia or phastosmia. Patients who have reported parosmia or phantosmia will be asked to complete a second part with six questions focusing on the quality of their olfactory distortion.
The abridged version of the Questionnaire of Olfactory Disorders - Negative Statements (sQOD-NS) | Measurement will be taken at time zero (pre-intervention) and 12 weeks (post-intervention)
  The sQOD-NS is a validated questionnaire that measures the quality of life specific to olfactory functions. The questionnaire measures 7 items with a 4-point Likert scale.

SECONDARY OUTCOMES:
Nasal Obstruction Symptom Evaluation (NOSE) | Measurement will be taken at time zero (pre-intervention)
  A visual analog scale (scale from "not a problem" to "severe problem") is used by participants to assess their nasal obstruction. The duration of this test is approximately 2 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes A Frasnelli, PhD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada